CLINICAL TRIAL: NCT01150539
Title: Effects of Physical Activity on Insulin Resistance and Adiposity in Polycystic Ovary Syndrome "Poly"
Brief Title: Effects of Exercise for Overweight Women With Polycystic Ovary Syndrome
Acronym: POLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Leanne Redman, Assistant Professor, Pennington Biomedical Research Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PBRC 26038
Record Dates: First submitted 2010-06-22; First posted 2010-06-25 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Polycystic Ovary Syndrome; Obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overweight/obese women with PCOS (Experimental): 10 overweight/obese women with polycystic ovary syndrome
  Interventions: Other: 16-week exercise training program; Other: Control Group without PCOS

INTERVENTIONS:
Other: 16-week exercise training program — The primary objective of the study is to investigate the effects of a 16-week exercise training program on insulin resistance and adiposity in overweight/obese women with PCOS.
Other: Control Group without PCOS — A group of overweight/obese women without PCOS will be enrolled as a control group and will be studied only once at baseline to allow for comparisons between the two study populations.

SUMMARY:
The effects of a 16-week exercise training program on insulin resistance and adiposity in overweight/obese women with Polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
Young, overweight/obese women with PCOS along with age and BMI-matched healthy controls without PCOS will be enrolled in this study. Participants will have assessments of body composition (by DEXA), visceral and ectopic fat (by MR), ovarian parameters (follicle size and number, by MRI) insulin sensitivity (by euglycemic hyperinsulinemic clamp), interstitial lipolysis (by microdialysis), whole body lipolysis and glycolysis (by stable isotopes), aerobic fitness (by VO2max test) and a fat biopsy performed across two clinic visits (1 outpatient visit, and 1 overnight stay). Participants in the control group will undergo these assessments once only, whereas participants in the PCOS Group will have these assessments twice, once at baseline and once following a 16 week supervised aerobic exercise program. Throughout the exercise program body weight will be measured weekly and menstrual cycle frequency will be documented on a calendar. Additionally, vital signs, weight, waist and hip circumferences will be measured and a fasting blood sample collected every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-30, inclusive.
* BMI greater than or equal to 25.
* Sedentary lifestyle - not currently exercising more than 60 minutes per week.
* A medical diagnosis of polycystic ovary syndrome. The diagnosis will be compared with the most recent international criteria1. Together with irregular menses (fewer than 6 cycles per year), participants must also have at least one of the following characteristics;

  1. presence of polycystic ovaries on transvaginal ultrasound, >10 cysts, 2-8 mm in diameter (ultrasound will not be done in this study however; ultrasound reports will be used if available) and/or
  2. clinical manifestations (hirsutism) examined by the PI at the screening visit or biochemical evidence (elevated testosterone or free androgen index) of hyperandrogenism, determined by fasting blood sample collected during the screening visit.
* Women enrolling for the non-PCOS control group are required to have regular menstrual cycles (one cycle per month).

Exclusion Criteria:

* Individuals with a history of cardiovascular disease or an elevated blood pressure above 160/90 mmHg.
* Individuals with a history of Diabetes (Type 1 or Type 2).
* Individuals with a history of Kidney, Liver or Heart disease.
* Individuals with untreated thyroid disease.
* Individuals who smoke.
* Individuals who exercise more than 60 minutes per week.
* Individuals who use medications including contraceptives (medications used to treat thyroid disease are permitted).
* Individuals with alcoholism or other substance abuse.
* Individuals who are pregnant or lactating (breast feeding).
* Individuals who become pregnant throughout the study will be excluded.
* Individuals who are trying to become pregnant.
* Control subjects will be excluded if they have irregular menses (fewer than 1 cycle per month).
* Unable to complete approximately 60 minutes of medium intensity exercise per day (5 days per week) at the Pennington Health and Fitness Center (PCOS Group Only).

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2007-01; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change in Insulin sensitivity as measured by the euglycemic hyperinsulinemic clamp | Baseline and 16-weeks
  16-weeks of aerobic exercise training on: peripheral insulin sensitivity (euglycemic-hyperinsulinemic clamp) and catecholamines (microdialysis) during a euglycemic-hyperinsulinemic clamp.

SECONDARY OUTCOMES:
Change in adiposity (whole body measurement by dual x-ray absorptiometry and visceral measured by magnetic resonance imaging) | Baseline and 16-weeks
  16-weeks of aerobic exercise training on total and free testosterone concentraions and frequency of menstruation, Body lipolysis, and visceral fat.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Readman, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States